CLINICAL TRIAL: NCT07263139
Title: A Phase 2a Trial to Investigate Safety, Tolerability and Exploratory Clinical Efficacy of AGP100 in Patients With Catecholaminergic Polymorphic Ventricular Tachycardia (PACE-CPVT)
Brief Title: Safety, Tolerability, and Exploratory Efficacy of AGP100 in Patients With Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agiana Pharmaceuticals (Industry)
Collaborators: Link Medical Research AS (Unknown); Viedoc Technologies AB (Unknown); Vitas AS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGP100-C01; 2025-521611-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia
MeSH Terms: conditions — Polymorphic Catecholaminergic Ventricular Tachycardia

STUDY DESIGN:
Masking Description: There is no masking as the study is a single-arm, open-label study. It is an intra-patient dose escalation study where patients first receive a low dose of the drug, then an medium dose, and then a high dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AGP100 (Experimental): Within this single arm, three doses levels are planned in an intra-patient dose-escalation design. These will be administered in sequential treatment periods:
  * Daily dose of 5 mg (1 x 5 mg capsule), oral route, for a planned duration of 13 days (starting dose)
  * Daily dose of 25 mg (1 x 25 mg capsule), oral route, for a planned duration of 13 days
  * Daily dose of 50 mg (2 x 25 mg capsules), oral route, for a planned duration of 13 days
  Interventions: Drug: AGP100

INTERVENTIONS:
Drug: AGP100 — AGP100 is a capsule for oral administration. The drug substance is formulated as an encapsulated dry powder blend composed of 5 mg or 25 mg active ingredient and inactive excipients filled into a white, opaque, size 3 hard gelatine capsule. The drug product is a white to light brown solid, with low solubility in water.
  During study visits, participants will take IMP under supervision of the study staff. Participants will receive with the oral dose together with water. During the rest of each treatment period, participants will self-administer the IMP. Doses should be taken with water, as needed. Participants are to continue to take the IMP once per day until they attend the study visit that starts the next treatment period/the end of study visit.

SUMMARY:
This trial is conducted in patients with an inherited heart rhythm disorder called catecholaminergic polymorphic ventricular tachycardia (CPVT). This condition causes the heart to beat dangerously fast during situations of physical or emotional stress. CPVT is a serious condition that can limit the length and quality of patients' lives. Current treatment does not always prevent the abnormal heart rhythms that can occur as part of CPVT during strenuous exercise or stress, so new and improved medications are needed.

The main questions that the trial will answer are:

* How safe and tolerable is the drug AGP100; i.e, what medical problems do patients experience when taking the drug?
* Does the drug help CPVT patients to maintain a normal heart rhythm while they are exercising?
* How does the drug affect the levels of key heart cell signalling molecules?

Patients with a diagnosis of CPVT who are aged between 18 and 75 and experience abnormal heart rhythms during exercise, despite taking a stable dose of the medication(s) prescribed by their doctor for their CPVT can take part in this trial. Participants should have normal kidney and liver function and not have high blood pressure or a diagnosis of structural heart disease. Women who are pregnant or breastfeeding cannot take part in the study. Participants who may become pregnant (and their partners) need to use highly effective methods of contraception during the study and for 90 days after the study ends.

Participants will take part in the study for ten weeks. During this time, participants will be asked to take three different doses of the the drug (AGP100), as well as their normal heart medication. The drug is an oral capsule and each different dose will be taken once a day for 13 days. The study starts with participants taking a low dose for 2 weeks, then a medium dose and then a high dose. At each dose, participants will undergo a clinical examination, report any potential side effects and the treating doctor will investigate the safety, tolerability and side effects of AGP100. In total, participants will take AGP100 once a day for about six weeks. The last four weeks of the study will be a follow-up period where participants will not take AGP100.

During the study, participants will need to visit the hospital six times. The visits will be three outpatient appointments and three overnight stays.

DETAILED DESCRIPTION:
The investigational medicinal product (IMP) used in this study is AGP100, a selective small molecule inhibitor of phosphodiesterase 2 (PDE2) under development by Agiana Pharmaceuticals (the Sponsor) for the treatment of catecholaminergic polymorphic ventricular tachycardia (CPVT) and cardiac arrhythmias (abnormal heart rhythms) that occur in other cardiovascular diseases.

The clinical data generated to date support the continued development of AGP100, and non-clinical data held by the Sponsor provide evidence that inhibition of PDE2 can attenuate cardiac calcium overload arrhythmias. Together, this supports the development of AGP100, a specific PDE2 inhibitor, as the first member of a new class of antiarrhythmic therapies. AGP100 was well tolerated, with no safety signals observed during administration to 95 individuals at single doses up to 125 mg and multiple doses up to 75 mg. The formulation of AGP100 planned to be used in this study (oral capsules containing either 5 or 25 mg AGP100), has been previously administered, as has a similar dosing regimen.

This phase IIa study will evaluate safety, tolerability, and preliminary clinical efficacy of multiple ascending doses of AGP100 in participants with confirmed CPVT - i.e., a trial population within the proposed indication for AGP100, and will be the first study in which AGP100 has been administered to patients (rather than healthy volunteers).

Current first-line prophylactic treatment for CPVT is full-dose non-selective β-blockers, with the addition of flecainide as a second-line treatment in some patients. However, despite currently available therapies, significant unmet medical need exists due to adverse effects, drug interactions, and/or limited efficacy in maintaining normal heart rhythm on current standard of care therapy when the patients undergoes surges of adrenergic stimulation. Therefore, the objective of this phase IIa clinical study is to assess the safety and tolerability of increasing doses of AGP100 in CPVT patients and to obtain preliminary efficacy data to support the development of AGP100 as the first member of a new class of antiarrhythmic therapies for the treatment of CPVT and other cardiac arrhythmias.

AGP100 will be given together with current standard of care. As discussed above, non-clinical data suggests that positive synergy between β-blockers and AGP100 may be expected as they function through distinct, complimentary modes of action.

The dose levels to be evaluated are 5 mg once daily, 25 mg once daily, and 50 mg once daily, respectively. This study will use an intra-patient dose escalation design. As CPVT is an orphan disease and due to the small number of patients available, the study is single-arm and open-label. With the current trial design participants will serve as their own control using baseline data. The study aims to generate reliable initial data on the use of AGP100 in CPVT patients through qualitative analysis of safety, tolerability and efficacy data (e.g., exercise testing results, pharmacodynamic parameters), in order to establish proof-of-principle and inform the design of future clinical studies.

The study population will consist of male and female participants aged 18 to 75 years (inclusive) diagnosed with CPVT. A total of 10 participants is planned to be enrolled at a single study site. A sentinel dosing approach will be applied, where the first 2 participants will be enrolled and complete the study sequentially (one at a time). After completion of the study by the first 2 sentinel participants (without safety issues, as determined by the safety review committee [SRC]) the remaining participants will be enrolled and treated.

Participants will be selected based on a history of residual ectopy on exercise testing. Each potentially eligible participant will undergo exercise testing as part of the Screening assessments (prior to enrolment) to confirm eligibility and establish study-specific individual baseline parameters whilst on their current standard of care medication(s). Participants with residual ectopy on exercise testing at Screening will be included in the study. At Visit 2, participants will be admitted to the study site, have blood samples drawn and receive the first dose of once daily oral AGP100 (5 mg), starting the first 2-week (13-day) treatment period. AGP100 will be taken daily alongside the patient's standard of care medication. An exercise test will be performed 2 hours after dosing of IMP to assess safety and efficacy parameters. Participants will undergo 24-hour ECG monitoring (telemetry) while admitted to the study site and will be discharged the following day.

During the remainder of this, and each subsequent treatment period, participants will self-report taking each dose of AGP100 daily using an electronic patient reported outcomes (ePRO) system, available via their smartphone, tablet, or computer.

The day following the last dose of the first treatment period (Day 14), participants will be admitted to the study site overnight. During this visit, participants will have blood samples drawn and if the previous dose level is well tolerated, and it is deemed appropriate by the Investigator, the dose will be escalated to 25 mg AGP100 once daily for a second 2-week (13-day) treatment period. An exercise test will be performed 2 hours after dose-escalation to assess safety and efficacy parameters. Participants will undergo 24-hour ECG monitoring (telemetry) while admitted to the study site and will be discharged the following day.

The day following the last dose of the second treatment period (Day 27), participants will attend and be admitted to the study site overnight. During this visit, participants will have blood samples drawn and if the previous dose level is well tolerated and it is deemed appropriate by the Investigator, the dose will be escalated to 50 mg AGP100 once daily for a third 2-week (13-day) treatment period. An exercise test will be performed 2 hours after dose escalation. Participants will undergo 24-hour ECG monitoring (telemetry) while admitted to the study site and will be discharged the following day.

On the last day of the third treatment period (Day 39, end of treatment [EoT]), participants will attend the study site as outpatients. During this visit, participants will self-administer their final dose of AGP100, will have blood samples drawn, and undergo an exercise test 2 hours after the dose of AGP100. Participants will then enter a 4-week (28-day) follow-up period without any study treatment.

At the end of the follow-up period participants will attend the study site and a final exercise test will be performed (end of study [EoS]).

The total study duration for each participant will be 68 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures
2. Male or female, aged between 18 and 75 years (inclusive)
3. Clinical diagnosis of CPVT based on proven RYR2 mutation AND reproducible premature ventricular contraction with exercise or polymorphic or bidirectional ventricular tachycardia with exercise
4. Able and willing to undergo exercise testing (bicycle test) AND exhibits exercise-induced ventricular ectopic beats at Screening (at least 1 point on the VA scale)
5. On stable, maximum tolerated, dose of non-selective β-blocker for at least 4 weeks before Visit 1. The dosage and choice of β-blocker are to be determined by the patients' physician(s) before entry into the study and must remain unchanged throughout the conduct of the study. Participants taking a stable dose of flecainide for at least 4 weeks, in addition to β-blocker, are also eligible.
6. Clinical laboratory evaluations including clinical chemistry, haematology, urinalysis, thyroid function (including thyroid stimulating hormone, triiodothyronine, thyroxine, and free T4) and coagulation testing (activated partial thromboplastin time, and international normalized ratio) within the reference range, unless deemed not clinically significant by the Investigator
7. Willing to refrain from strenuous or new exercise for 24 hours before each study visit
8. Women of childbearing potential (WOCBP) agree to implement accepted and highly effective means of contraception from study entry until at least 33 days after study drug discontinuation (as per the Clinical Trials Facilitation and Coordination Group guidelines).

The main exclusion criteria are:

1. Diagnosis of structural heart disease, including coronary artery disease or heart failure with reduced ejection fraction (left ventricular ejection fraction <45%)
2. Participants who have had arrhythmias causing hemodynamic instability at previous exercise tests (performed while on the current standard of care treatment)
3. Participants having a sustained VT (VA score of 5) during the exercise tests performed as part of the screening activities
4. Participation in another clinical study with an investigational product or device within 60 days of 5 half-lives prior to Baseline (whichever is longer)
5. Medical history of severe anaphylactic reactions to any component(s) of the IMP
6. Sensitivity to any of the study treatments, or components thereof, or any drug or other allergy that, in the opinion of the Investigator precludes participation in the study
7. Hypersensitivity or contraindication to PDE2 inhibitor drugs
8. Use of PDE3, PDE4, or PDE5 inhibitor drugs.
9. Participants taking any antiarrhythmic drug(s) except flecainide and non-selective β-blockers
10. Significant hypertension (defined as systolic blood pressure of >160 mmHg and/or diastolic blood pressure of >95 mmHg). If the blood pressure results are out of range at Screening, the measurements can be repeated on the same day more than once, or at another convenient visit
11. Prolonged PR and/or QTc interval at Screening, defined as PR >240 ms or QTc >480 ms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From Day 1 (start of treatment) through Day 68 [EoS])
Changes in heart rate (HR) | Day 1, Day 2, Day 14, Day 15, Day 27, Day 28, Day 39 (End of Treatment), and Day 68 (EoS)
  Unit: beats per minute (bpm)
Changes in 12-lead electrocardiogram parameters: estimated ventricular frequency | Day 1, Day 2, Day 14, Day 15, Day 27, Day 28, Day 39 (End of Treatment), and Day 68 (EoS)
  Unit: bpm
Changes in 12-lead electrocardiogram parameters: PR | Day 1, Day 2, Day 14, Day 15, Day 27, Day 28, Day 39 (End of Treatment), and Day 68 (EoS)
  Unit: milliseconds (ms)
Changes in 12-lead electrocardiogram parameters: QRS | Day 1, Day 2, Day 14, Day 15, Day 27, Day 28, Day 39 (End of Treatment), and Day 68 (EoS)
  Unit: milliseconds (ms)
Changes in 12-lead electrocardiogram parameters: QTc | Day 1, Day 2, Day 14, Day 15, Day 27, Day 28, Day 39 (End of Treatment), and Day 68 (EoS)
  Unit: milliseconds (ms)
Tolerability of the IMP | From Day 1 (start of treatment) through Day 68 [EoS])
  This will be assessed as a binary parameter (tolerable Yes or No): If any of following changes in IMP dosing is deemed necessary, the participant will be classified as 'No':
  * Dose adjustments prescribed by the Investigator
  * Dose interruptions prescribed by the Investigator
  * Discontinuation of treatment

SECONDARY OUTCOMES:
Change from baseline in the amount and complexity of exercise-induced ventricular ectopic beats as assessed using the ventricular arrythmia (VA) score | Day 1 (post-dose), Day 14, Day 27, Day 39, and Day 68
  The VA score is reported as an ordinal value on a scale from 0 to 5. 0 = no inducible VA, 1 = isolated inducible premature ventricular contractions (PVCs); <10 beats per minute, 2 = bigeminal PVCs and/or frequent PVCs (≥10 per minute), 3 = ventricular couplet, 4 = non-sustained ventricular tachycardia (VT) (≥3 consecutive PVCs at a rate of >100 beats per minute [bpm], terminating spontaneously), 5 = sustained VT (≥30 seconds and rate >100 bpm) or ventricular fibrillation
Change from baseline in urine cyclic guanosine monophosphate (cGMP) levels | Day 1 (post-dose), Day 14, Day 27, Day 39, and Day 68
Change from baseline in urine cyclic adenosine monophosphate (cAMP) levels | Day 1 (post-dose), Day 14, Day 27, Day 39, and Day 68
Change from baseline in plasma cGMP levels | Day 1 (post-dose), Day 14, Day 27, Day 39, and Day 68
Change from baseline in plasma cAMP levels | Day 1 (post-dose), Day 14, Day 27, Day 39, and Day 68

CONTACTS AND LOCATIONS:
Overall Officials: Rizwan Hussain, MD PhD, Study Director — Agiana Pharmaceuticals AS
Locations (1):
- Department of Cardiology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.